CLINICAL TRIAL: NCT01035112
Title: Magnetic Resonance Imaging of Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-10748; 13IB-0074 (Other: NIH); 75763 (Other: Stanford IRB (old)); R01CA249893 (NIH); BRSNSTU0004 (Other: OnCore); NCI-2024-01929 (Registry Identifier: NCI-Clinical Trials Reporting Program)
Record Dates: First submitted 2009-12-17; First posted 2009-12-18 (Estimated); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer; Breast Cancer Non-invasive Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Magnetic Resonance Imaging (MRI) of Breast Cancer (Experimental): Contrast-enhanced magnetic resonance imaging (MRI) using the standard department of Radiology MRI screening procedures. The duration of scanning may be variable, but will not exceed 90 minutes.
  Interventions: Procedure: MRI

INTERVENTIONS:
Procedure: MRI

SUMMARY:
To compare magnetic resonance imaging (MRI) with more well established diagnostic imaging techniques to determine which method best finds and defines breast cancer.

ELIGIBILITY:
INCLUSION CRITERIA

* Female
* Documented breast physical examination,
* Documented mammography within 3 months of the MR studies
* Palpable or mammographically-detected suspect breast lesions
* Women who have already undergone lumpectomy for breast cancer and have post-biopsy/post-radiation changes will be eligible if they have mammographically-detected or palpable breast abnormalities which are sufficiently suspicious to merit core needle or surgical biopsy.

EXCLUSION CRITERIA:

* Male by birth
* Able to complete the MR examination. Subjects will be interviewed by one of the investigators for the usual contraindications to
* MR contraindications including
* Pacemakers
* Metallic implants
* Severe claustrophobia
* Aneurysm clips
* Pregnancy
* Current lactation
* Other conditions precluding proximity to a strong magnetic field.
* Received an enhanced MR procedure within 48 hours,
* Iodinated contrast within six hours,
* Known sensitivity to MR contrast agents,
* Not likely to complete the study in full or
* Other clinical reason which would preclude participation in the protocol.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — female by birth
Enrollment: 500 (Estimated)
Dates: Start 1995-04-01 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
To compare magnetic resonance imaging (MRI) with more well established diagnostic imaging techniques to determine which method best finds and defines breast cancer. | Length of one MRI scan

CONTACTS AND LOCATIONS:
Overall Officials: Bruce L Daniel, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No